CLINICAL TRIAL: NCT06747988
Title: Prospective Study Evaluating the Use of a Novel Through - the- Scope Suturing System as a Dynamic Traction Device During ESD: A Feasibility Study
Brief Title: Feasibility and Prospective Study of a Dynamic Traction Device for Use During ESD
Status: Not yet recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Salmaan Azam Jawaid, MD, Assistant professor of Medicine, Baylor College of Medicine
Other Study IDs: H-56820
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Gastrointestinal Neoplasms
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Traction Device — After circumferential incision and trimming the submucosa at the incision's edge, dissection is initiated until approximately 20 to 30% of the anal side (for colonic lesions) or oral side (for gastric lesions) of lesion has been dissected leaving a flap of at least 1 cm in length. Once the mucosal flap is created the X-tack device is introduced through the endoscope channel. The first tack is placed on the opposite wall of the lesion, the 2nd and 3rd tack will then be placed next to each other on the mucosal flap portion of the lesion. The 4th tack does not have to be placed but can be used to generate further traction at any time. Clips can be placed along the suture and clipped to the wall at any point to change angulation of traction. The sutures can then be cut and released from the tissue

SUMMARY:
The goal of this prospective study at Baylor St. Luke's Medical Center is to investigate the the efficacy and safety of using the novel TTS helix tack suture device as a dynamic traction device during colon and gastric endoscopic submucosal dissection (ESD). The investigators of this study hypothesize that a dynamic traction during ESD can be less traumatic than with other traction devices.

DETAILED DESCRIPTION:
Endoscopic submucosal dissection (ESD) is the mainstay of treatment for complex gastrointestinal polyps, particularly those with a higher risk of superficial submucosal invasion. To facilitate endoscopic dissection, traction is frequently used, particularly in tough locations or when fibrosis is present [1]. Traction assisted ESD is particularly attractive when other techniques, such as tunneling or pocket formation, are not effective.

Tissue traction can be applied by several methods including gravity, mucosal tension, water pressure, and adjusting the patient's body position [2]. Additionally, traction can also be applied using devices such as clip and line, snare, band assisted or using dedicated over-the-scope devices, which can be cumbersome and costly. Despite multiple publications about the efficacy of traction devices in the East, there are few published data from the West [3]. Furthermore, an easy to use through the scope (TTS) dynamic traction device has yet to be developed. Recently, a novel TTS helix tack and suture device (X-tack, Apollo Endosurgery, Austin, Tex, USA) was FDA approved to help facilitate closure of post-resection defects [4]. However, clinical experience suggests the tack and suture system can also be used as a form of dynamic traction during ESD, similar to effective techniques using traditional suture-pulley systems for countertraction during ESD [5]. The traditional suture-pulley system, however, can be cumbersome to assemble as multiple parts are needed to configure it appropriately [6]. Additionally, attaching the suture to the designated areas requires use of multiple costly clips and if repositioning is needed, removal of the clip can be traumatic to the tissue. With the novel TTS suture system (X-tack), four tacks are already assembled along one suture line, thus a suture-pulley countertraction system can be employed without having to assemble multiple parts. In addition, the degree and angulation of traction can be altered simply by pulling, releasing or even redirecting the suture towards a different axis, supporting a dynamic traction during ESD. Finally, removal of the tack, if required, can be less traumatic than with other traction devices. Despite its potential advantages, use of X-tack as countertraction pulley system during ESD has not been formally studied. We looked to investigate the efficacy and safety of using the novel TTS helix tack suture device as a dynamic traction device during colon and gastric ESD.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥ 18 years old.
2. Patients can provide informed consent.
3. The patient is referred for ESD procedure of colonic or gastric neoplastic lesions and with one of the following criteria:

A- Lesions with prior failed resection of any size. B- Granular lateral spreading tumors (GLST) more than 30 mm. C- Non granular lateral spreading tumors (NGLST) more than 20 mm. D- Any lesion with suspected superficial submucosal invasion. E- Subepithelial lesions.

Exclusion Criteria:

1. The patient is < 18 years old.
2. The patient refuses and/or is unable to provide consent.
3. The patient is a pregnant woman.
4. Lesions with morphology: pedunculated type (Paris Ip, Ips).
5. Appendiceal orifice or IC valve lesions
6. Patients with lesions removed with other techniques besides ESD (submucosal tunneling technique [STER] or EMR).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ESD procedure at Baylor St. Luke's Medical Center - Houston, TX.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Technical success | Day 1 (procedure day)
  Being able to dissect the lesion to facilitate en bloc removal (removal of the entire tumor endoscopically in one piece)

SECONDARY OUTCOMES:
Dissection speed | Day 1 (procedure day)
  Length of time to perform endoscopic submucosal dissection by the operator as measured by calculating area of lesion divided by time (cm^2/hours).
R0 and curative resection rates | Day 1 (procedure day)
  As collected
Total procedure time | Day 1 (procedure day)
  Total procedure time to perform ESD from scope in to scope out
NASA Task Load Index | Day 1 (procedure day)
  Method assesses work load on five 7-point scales. Increments of high, medium and low
Intraprocedural adverse events | Day 1 (procedure day), up to 48 hours after procedure.
  Such as musclaris propria injury and bleeding (related to or not related to the traction devices).
Post-procedural adverse events | 1 month post-procedure
  As reported per subject follow-ups with the patient within 1 month.
Abdominal pain | 1 hour post-procedure, 24 hours post-procedure.
  Collected at 1 hour and 24 hours after procedure utilizing the Visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no expected significant increased risk associated with the use of the traction device in ESD beyond what the current standard is for the procedure. Loss of confidentiality is the only other risk associated with this project. All measures to ensure patient confidentiality will be employed. Data will be coded and entered into a password-protected computer. Only the Principal Investigator and Study Research Coordinators will have access to data with patient identifiers. There will be no disclosure of a patients protected health information. Paper copies of the study documents will be created only as needed and only shown to the investigators listed in the study. Once the study is completed, all paper copies will be destroyed. If the results of the study are published or used in any presentations, all patient related information will be coded.

REFERENCES:
- [Result] Tanaka S, Terasaki M, Kanao H, Oka S, Chayama K. Current status and future perspectives of endoscopic submucosal dissection for colorectal tumors. Dig Endosc. 2012 May;24 Suppl 1:73-9. doi: 10.1111/j.1443-1661.2012.01252.x. PMID 22533757
- [Result] Othman MO, Jawaid SA, Rungta M, Sur N, Dhingra S. Double-balloon endolumenal intervention platform with flexible grasper to expedite colonic endoscopic submucosal dissection. VideoGIE. 2020 Dec 26;6(3):144-146. doi: 10.1016/j.vgie.2020.11.014. eCollection 2021 Mar. No abstract available. PMID 33738368
- [Result] Nagata M. Usefulness of underwater endoscopic submucosal dissection in saline solution with a monopolar knife for colorectal tumors (with videos). Gastrointest Endosc. 2018 May;87(5):1345-1353. doi: 10.1016/j.gie.2017.11.032. Epub 2017 Dec 12. PMID 29242059
- [Result] Hernandez A, Marya NB, Sawas T, Rajan E, Gades NM, Wong Kee Song LM, Abu Dayyeh BK, Buttar N, Storm AC. Gastrointestinal defect closure using a novel through-the-scope helix tack and suture device compared to endoscopic clips in a survival porcine model (with video). Endosc Int Open. 2021 Apr;9(4):E572-E577. doi: 10.1055/a-1370-9256. Epub 2021 Apr 12. PMID 33860074
- [Result] Ge PS, Thompson CC, Jirapinyo P, Aihara H. Suture pulley countertraction method reduces procedure time and technical demand of endoscopic submucosal dissection among novice endoscopists learning endoscopic submucosal dissection: a prospective randomized ex vivo study. Gastrointest Endosc. 2019 Jan;89(1):177-184. doi: 10.1016/j.gie.2018.08.032. Epub 2018 Aug 25. PMID 30148993
- [Result] Rieder E, Makris KI, Martinec DV, Swanstrom LL. The suture-pulley method for endolumenal triangulation in endoscopic submucosal dissection. Endoscopy. 2011;43 Suppl 2 UCTN:E319-20. doi: 10.1055/s-0030-1256774. Epub 2011 Oct 21. No abstract available. PMID 22020705
- [Result] Burgess NG, Bassan MS, McLeod D, Williams SJ, Byth K, Bourke MJ. Deep mural injury and perforation after colonic endoscopic mucosal resection: a new classification and analysis of risk factors. Gut. 2017 Oct;66(10):1779-1789. doi: 10.1136/gutjnl-2015-309848. Epub 2016 Jul 27. PMID 27464708